CLINICAL TRIAL: NCT00944385
Title: Effects of Ulinastatin on Myocardial Protection and Blood Loss in Patients Undergoing Aortic Valve Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Young Lan Kwak/ Professor, MD, Severance Hospital
Other Study IDs: 4-2009-0079
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Abnormal Aortic Valve
MeSH Terms: interventions — urinastatin

ARMS (2):
- ulinastatin (Experimental): Administer with 30,000U /ulinastatin
  Interventions: Drug: ulinastatin
- C group (Placebo Comparator): administer normal saline
  Interventions: Drug: ulinastatin

INTERVENTIONS:
Drug: ulinastatin — Administer 30000U/ulinastatin. Comparison of different dosages of drug.

SUMMARY:
According to TEG (thromboelastography), as maximum amplitude is increased the amount of bleeding and transfusion and Cardiac enzyme is reduced by using ulinastatin.

ELIGIBILITY:
Inclusion Criteria:

* 40% below of output of left ventricle
* tricuspid valve failure from moderate to severe
* urgent surgery required
* infectious endocarditis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Younglan Kwak, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea